CLINICAL TRIAL: NCT03128047
Title: HUMC 1612: A Phase I Trial of the Optune NovoTTF-200A System With Concomitant Temozolomide and Bevacizumab in Pediatric Patients With High-grade Glioma
Brief Title: HUMC 1612: Optune NovoTTF-200A System
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hackensack Meridian Health (Other)
Collaborators: NovoCure Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro2016-0583
Record Dates: First submitted 2017-01-05; First posted 2017-04-25 (Actual); Results first posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: High Grade Glioma; Ependymoma
Keywords: pediatric cancer; brain tumor; glioblastoma; high grade brain tumor; malignant brain tumor; recurrent brain tumor
MeSH Terms: conditions — Glioma; Ependymoma; Neoplasms; Brain Neoplasms; Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Recurrent high grade gliomas and ependymomas (Experimental): Recurrent high-grade glioma and ependamoma patients will receive treatment with the Optune NovoTTF-200A system as monotherapy.
  Interventions: Device: Optune NovoTTF-200A System Optune NovoTTF-200A System receive treatment with 200kHz for a minimum of 18 hours per day in 28 day cycles combined with Temozolomide and Bevacizumab.
  Interventions: Device: Optune NovoTTF-200A System

INTERVENTIONS:
Device: Optune NovoTTF-200A System — Optune NovoTTF-200A System receive treatment with 200kHz for a minimum of 18 hours per day in 28 day cycles combined with Temozolomide and Bevacizumab.

SUMMARY:
The purpose of this study is to determine if the Optune NovoTTF-200A device can be safely used in combination with chemotherapy in pediatric patients with recurrent high-grade glioma and ependemoma.

DETAILED DESCRIPTION:
This phase I trial will utilize a standard 3+3 design to determine the safety and tolerability of the Optune NovoTTF-200A System in pediatric patients with recurrent high-grade glioma end ependemomas.

Patients will receive treatment with the Optune NovoTTF-200A System along with Temozolomide and Bevacizumab and will consist of children with recurrent high-grade gliomas and Ependamomas. Patients enrolled will receive treatment with the Optune NovoTTF-200A with 200kHz for a minimum of 18 hours per day in 28 day cycles as monotherapy. Phase I safety evaluation will take place over the initial two cycles (56 days) of treatment. Following the completion of the safety evaluation period, patients will continue to receive treatment in 28 day cycles, which may be repeated continuously without therapy interruption for 12 cycles or until clinical criteria for discontinuation are met. Patients how appear to benefit from this treatment may be allowed to continue treatment beyond 12 cycles if approved by the study Principle Investigator.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a minimum head circumference of 44 cm
* Patients must have a histologically- or cytologically-confirmed supratentorial high-grade glioma or supratentorial ependemoma.
* Patients with metastatic disease involving the infratentorium or spinal cord are eligible providing that they have a supratentorial tumor that is able to be targeted with TTFields.
* Eligible pathologic diagnoses include:

High-grade Glioma (WHO Grade III or IV): Anaplastic Astrocytoma, Astroblastoma, Diffuse Midline Glioma, Glioblastoma, Gliosarcoma Ependymoma (WHO Grade II or III):Ependymoma, Anaplastic Ependymoma

* Patients with high-grade glioma must must have be newly-diagnosed or have a tumor that is progressive or recurrent following standard treatment. Patients with ependymoma must have a tumor that is progressive or recurrent following standard treatment.
* Patients must have received the maximal feasible resection of their tumor and radiation therapy (unless contraindicated due to patient age) as part of their initial treatment prior to study enrollment.
* Patients must be enrolled before treatment begins. Treatment must start within 14 days of study enrollment.
* All clinical and laboratory studies to determine eligibility must be performed within 7 days prior to enrollment unless otherwise indicated in the eligibility section.
* Newly-diagnosed patients must begin therapy within six weeks of the completion of radiotherapy, or within six weeks of surgical resection if radiotherapy is contraindicated.
* Recurrent high-grade glioma patients must begin therapy within four weeks of documented tumor progression by MRI scan.
* Patients must have a Lansky or Karnofsky performance status score of ≥ 50%, corresponding to ECOG categories of 0, 1 or 2. Use Karnofsky for patients > 16 years of age and Lansky for patients ≤ 16 years of age. Patients who are unable to walk because of paralysis, but who are up in a wheelchair will be considered ambulatory for the purpose of assessing the performance score.
* Able to undergo adequate tumor imaging, via magnetic resonance imaging (MRI) scan to evaluate disease evolution.
* Adequate hematologic, renal, liver function as demonstrated by laboratory values: ANC ≥ 1,000/ul Hemoglobin ≥8.0 gm/dl Platelet count ≥ 100,000/ul

Adequate Liver Function Defined As:

* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) for age, and
* SGPT (ALT) < 2.5 x upper limit of normal (ULN) for age. Adequate Renal Function Defined As Either
* Creatinine clearance or radioisotope GFR ≥ 70ml/min/1.73m2
* or a serum creatinine less than or equal to the institutional normal for age

  * Negative pregnancy test in women of childbearing potential within 7 days of initiating investigational therapy
  * Recent mothers must agree not to breast feed while receiving medications on study
  * Patient or legal guardian must give written, informed consent or assent (when applicable).
  * Able to swallow and ingest oral medication or have a NG or G-tube for drug administration
  * Urine protein should be screened by urine analysis. If protein ≥ 2+ on urinalysis, then Urine Protein Creatinine (UPC) ratio should be calculated. If UPC ratio > 0.5, 24-hour urine protein should be obtained and the level should be < 1000 mg for patient enrollment.

Note: UPC ratio of spot urine is an estimation of the 24 urine protein excretion - a UPC ratio of 1 is roughly equivalent to a 24-hour urine protein of 1000 mg. UPC ratio is calculated using one of the following formula:

* [urine protein]/[urine creatinine] - if both protein and creatinine are reported in mg/dL
* [(urine protein) x0.088]/[urine creatinine] - if urine creatinine is reported in mmol/L
* Adequate Coagulation Defined As: PT/INR ≤ 1.5 x upper limit of normal

Exclusion Criteria:

* Age less than 5 or greater than or equal to 18 years
* Head circumference < 44 cm
* Absence of supratentorial tumor
* Use of any other investigational drug within five half-lives of that drug prior to the initiation of protocol therapy
* Anti-cancer therapy within 4 weeks prior to the initiation of protocol therapy (6 weeks for mitomycin and nitrosureas, 4 weeks for curative-intent radiotherapy, and 2 weeks for palliative radiotherapy)
* Any National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE version 4.0) >Grade 1 toxicities from prior chemotherapy or radiotherapy that could impact on safety outcome assessment
* Any surgery within 14 days prior to initiation of protocol therapy (excluding shunt or line insertion)
* Implanted pacemaker, programmable shunts, defibrillator, deep brain stimulator, other implanted electronic devices in the brain, or documented clinically significant arrhythmias.
* Evidence of increased intracranial pressure (midline shift > 5mm, clinically significant papilledema, vomiting and nausea or reduced level of consciousness) Patients receiving escalating doses of corticosteroids to control symptoms of increased intracranial pressure (e.g., require a stable or decreasing dose of corticosteroids for at least 7 days prior to enrollment) will also be excluded.
* Known > Grade 1 intracranial or intratumoral hemorrhage either by CT or MRI scan within the last 1 month. Patients with resolving hemorrhage changes, punctuate hemorrhage or hemosiderin may enter the study
* Pregnant female patients, Pregnancy tests with a negative result must be obtained in all post-menarchal females.
* Lactating females must agree they will not breastfeed a child while on this study.
* Males and females of reproductive potential may not participate unless they agree to use an effective contraceptive method and continue to do so for at least 6 months after the completion of therapy.
* Any serious and/or unstable pre-existing medical, psychiatric or other condition which in the Investigator's opinion could interfere with subject safety, obtaining written informed consent, or compliance with the study protocol
* Known hypersensitivity to temozolomide or bevacizumab
* Patients who are unable to take oral medications because of significant uncontrolled vomiting will be excluded.
* Patients must not have a history of myocardial infarction, severe or unstable angina, clinically significant peripheral vascular disease, Grade 2 or greater heart failure, or serious and inadequately controlled cardiac arrhythmia.
* Patients must not have a known clinically significant bleeding diathesis or coagulopathy
* Patients who have experienced arterial thromboembolic events, including transient ischemic attacks or cerebrovascular accidents are excluded from participation.
* Patients must not have been previously diagnosed with a deep venous thrombosis (including pulmonary embolism), and must not have a known thrombophilic condition (e.g., protein S, protein C, antithrombin III deficiency, Factor V Leiden or Factor II G202'0A mutation, homocysteinemia, or antiphospholipid antibody syndrome).
* Patients must not have a history of an abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within the last 6 months prior to study entry.
* Patients with a serious or non-healing wound, ulcer, or bone fracture are not eligible for this study.
* Patients with a history of allergic reaction to Chinese hamster ovary cell products, or other recombinant human antibodies are ineligible.

Ages: 5 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2025-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Derek Hanson, MD, Principal Investigator — Joseph M. Sanzari Children's Hospital at Hackensack University Medical Center
Locations (2):
- United States (2):
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Joseph M. Sanzari Children's Hospital at Hackensack University Medical Center, Hackensack, New Jersey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kirson ED, Gurvich Z, Schneiderman R, Dekel E, Itzhaki A, Wasserman Y, Schatzberger R, Palti Y. Disruption of cancer cell replication by alternating electric fields. Cancer Res. 2004 May 1;64(9):3288-95. doi: 10.1158/0008-5472.can-04-0083. PMID 15126372
- [Background] Kirson ED, Dbaly V, Tovarys F, Vymazal J, Soustiel JF, Itzhaki A, Mordechovich D, Steinberg-Shapira S, Gurvich Z, Schneiderman R, Wasserman Y, Salzberg M, Ryffel B, Goldsher D, Dekel E, Palti Y. Alternating electric fields arrest cell proliferation in animal tumor models and human brain tumors. Proc Natl Acad Sci U S A. 2007 Jun 12;104(24):10152-7. doi: 10.1073/pnas.0702916104. Epub 2007 Jun 5. PMID 17551011
- [Background] Stupp R, Taillibert S, Kanner AA, Kesari S, Steinberg DM, Toms SA, Taylor LP, Lieberman F, Silvani A, Fink KL, Barnett GH, Zhu JJ, Henson JW, Engelhard HH, Chen TC, Tran DD, Sroubek J, Tran ND, Hottinger AF, Landolfi J, Desai R, Caroli M, Kew Y, Honnorat J, Idbaih A, Kirson ED, Weinberg U, Palti Y, Hegi ME, Ram Z. Maintenance Therapy With Tumor-Treating Fields Plus Temozolomide vs Temozolomide Alone for Glioblastoma: A Randomized Clinical Trial. JAMA. 2015 Dec 15;314(23):2535-43. doi: 10.1001/jama.2015.16669. PMID 26670971
- [Background] Chaudhry A, Benson L, Varshaver M, Farber O, Weinberg U, Kirson E, Palti Y. NovoTTF-100A System (Tumor Treating Fields) transducer array layout planning for glioblastoma: a NovoTAL system user study. World J Surg Oncol. 2015 Nov 11;13:316. doi: 10.1186/s12957-015-0722-3. PMID 26558989

RESULTS

PARTICIPANT FLOW:
Groups:
- Recurrent High Grade Gliomas and Ependymomas: Recurrent high-grade glioma and ependamoma patients will receive treatment with the Optune NovoTTF-200A system as monotherapy.
  Interventions: Device: Optune NovoTTF-200A System Optune NovoTTF-200A System receive treatment with 200kHz for a minimum of 18 hours per day in 28 day cycles combined with Temozolomide and Bevacizumab.
  Optune NovoTTF-200A System: Optune NovoTTF-200A System receive treatment with 200kHz for a minimum of 18 hours per day in 28 day cycles combined with Temozolomide and Bevacizumab.
Period: Overall Study
Arm/Group | Recurrent High Grade Gliomas and Ependymomas
Started | 7
Completed | 6
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Recurrent High Grade Gliomas and Ependymomas
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 16.4 [13 to 21]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 3
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Safety of the Optune NovoTTF-200A System When Used Alone in Pediatric Patients With Recurrent High-grade Gliomas.
Description: Number of participants receiving treatment with the Optune NovoTTF-200A System with treatment-related adverse events as assessed by CTCAE v4.0.
Time Frame: 56 Days
Population: Number of patients with device related adverse events
Measure: Count of Participants; unit: Participants
Arm/Group | Recurrent High Grade Gliomas and Ependymomas
Number analyzed (Participants) | 6
Participants | 0

2. Primary Outcome: Tolerability of the Optune NovoTTF-200A System When Used Alone in Pediatric Patients With Recurrent High-grade Gliomas.
Description: Number of participants receiving treatment with the Optune NovoTTF-200A System with who return tolerability questionnaire and found the device tolerable
Time Frame: 56 Days
Population: Number of patients who found the device tolerable
Measure: Count of Participants; unit: Participants
Arm/Group | Recurrent High Grade Gliomas and Ependymomas
Number analyzed (Participants) | 6
Participants | 6

3. Secondary Outcome: Assess the Progression Free of Patients Treated on This Study Protocol to Aid in the Future Development of Pediatric Phase II/III Studies Using the Optune NovoTTF-200A System.
Description: Number of patients who are progression-free. Disease progression is defined as 25% or more increase in the product of perpendicular diameters of ANY target lesion, taking as reference the smallest product observed since the start of treatment (see exception below), OR the appearance of one or more new lesions, OR worsening neurologic status not explained by causes unrelated to tumor progression (e.g., anticonvulsant or corticosteroid toxicity, electrolyte disturbances, sepsis, hyperglycemia, presumed post-therapy swelling etc.) PLUS any increase in tumor cross-sectional area (or tumor volume).
Time Frame: Up to 2 years after study entry
Measure: Count of Participants; unit: Participants
Arm/Group | Recurrent High Grade Gliomas and Ependymomas
Number analyzed (Participants) | 6
Participants | 1

4. Secondary Outcome: Assess the Overall Survival of Patients Treated on This Study Protocol to Aid in the Future Development of Pediatric Phase II/III Studies Using the Optune NovoTTF-200A System.
Description: Number of patients who were alive at 2 years post study entry
Time Frame: Up to 2 years after study entry
Population: Number of patients who were alive at 2 years post study entry
Measure: Count of Participants; unit: Participants
Arm/Group | Recurrent High Grade Gliomas and Ependymomas
Number analyzed (Participants) | 6
Participants | 1

ADVERSE EVENTS:
Time Frame: For 30 days after participants stopped wearing the device, up to 2 years.
Arm/Group | Recurrent High Grade Gliomas and Ependymomas
All-Cause Mortality (participants affected / at risk) | 5/6
Serious Adverse Events (participants affected / at risk) | 3/6
Other Adverse Events (participants affected / at risk) | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recurrent High Grade Gliomas and Ependymomas (N=6)
Hypertension (Cardiac disorders) | 3 (6)
Proteinuria (Renal and urinary disorders) | 1 (1)
Allergic reaction to drug (Immune system disorders) | 1 (1)
Surgical site Wound (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2023-08-07): https://cdn.clinicaltrials.gov/large-docs/47/NCT03128047/Prot_000.pdf